CLINICAL TRIAL: NCT01147718
Title: An Open-label, Sequential Study to Evaluate the Pharmacokinetics of Digoxin When Coadministered With Albiglutide in Healthy Adult Subjects
Brief Title: A Drug Interaction Study of Albiglutide and Digoxin
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 111680
Record Dates: First submitted 2010-04-29; First posted 2010-06-22 (Estimated); Last update posted 2017-06-12 (Actual); Status verified 2017-06

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: pharmacokinetics; albiglutide; Healthy volunteer; digoxin
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Digoxin; rGLP-1 protein

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- digoxin plus albiglutide (Experimental): A single dose of 0.5mg digoxin administered on Day 1 followed by 5 weekly subcutaneous injections of albiglutide, followed by a further single dose of 0.5mg digoxin on Day 38.
  Interventions: Biological: digoxin plus albiglutide

INTERVENTIONS:
Biological: digoxin plus albiglutide — A single dose of 0.5mg digoxin on Day 1 followed by 5 weekly doses of subcutaneous albiglutide, followed by a single dose of 0.5mg digoxin on Day 38.

SUMMARY:
This Phase I, open-label, sequential, single-center study evaluates the pharmacokinetics of digoxin when coadministered with albiglutide in healthy adult subjects.

DETAILED DESCRIPTION:
This Phase I, open-label, sequential, single-center study evaluates the pharmacokinetics of digoxin when coadministered with albiglutide in healthy adult subjects. Subjects will receive a single dose of digoxin on Day 1 followed by 5 weekly subcutaneously injected doses of albiglutide and a second single dose of digoxin on Day 38. To determine the plasma pharmacokinetic parameters of digoxin after drug administration alone and after multiple doses of albiglutide, blood samples will be collected after each dose of digoxin.

ELIGIBILITY:
Inclusion Criteria:

* healthy volunteers
* female subjects must be of nonchildbearing potential
* no clinically significant diseases or clinically significant abnormal laboratory values
* body mass index (BMI) is >/=18 kg and ≤30 kg/m2
* a nonsmoker

Exclusion Criteria:

* positive test results for hepatitis B, hepatitis C or human immunodeficiency virus
* female subject is pregnant or breast-feeding
* history of any anaphylactic reaction to any drug
* history of significant cardiovascular or pulmonary dysfunction
* current or chronic history of liver disease
* history of alcohol or substance abuse
* history of thyroid disease or dysfunction
* history of gastrointestinal surgery or disease
* history of pancreatitis
* history of cholecystitis or other gallbladder disease
* previously received any GLP-1 mimetic compound (e.g., exenatide)

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2010-06-11 (Actual); Primary Completion 2010-11-29 (Actual); Study Completion 2010-11-29 (Actual)

PRIMARY OUTCOMES:
The pharmacokinetic parameters of digoxin with and without albiglutide | 38 days

SECONDARY OUTCOMES:
Safety of digoxin with and without albiglutide | 38 days

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Austin, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Background] Bush M, Scott R, Watanalumlerd P, Zhi H, Lewis E. Effects of multiple doses of albiglutide on the pharmacokinetics, pharmacodynamics, and safety of digoxin, warfarin, or a low-dose oral contraceptive. Postgrad Med. 2012 Nov;124(6):55-72. doi: 10.3810/pgm.2012.11.2613. PMID 23322139
- [Derived] Young MA, Wald JA, Matthews JE, Scott R, Hodge RJ, Zhi H, Reinhardt RR. Clinical pharmacology of albiglutide, a GLP-1 receptor agonist. Postgrad Med. 2014 Nov;126(7):84-97. doi: 10.3810/pgm.2014.11.2836. PMID 25387217
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- See also: Results for study 111680 can be found on the GSK Clinical Study Register. — https://gsk-clinicalstudyregister.com/study/111680?search=study&search_terms=111680#rs
- Available data/document: Clinical Study Report: 111680 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 111680 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 111680 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 111680 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 111680 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 111680 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 111680 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register